CLINICAL TRIAL: NCT06813521
Title: Evaluation of the Effect of a Lotion on Antidandruff and on Mediating Microbiome Rebalance Versus Vehicle and Reference on Volunteers
Brief Title: Antidandruff Lotion Mediating Microbiome Rebalance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACR-PAN1-19-01989
Record Dates: First submitted 2024-11-12; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Dandruff
Keywords: lotion; antidandruff; microbiome rebalance
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Intervention Model Description: cosmetic product
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NaP1%+VitCG3% leave-on lotion (Experimental)
  Interventions: Other: NaP1%+VitCG3% leave-on lotion (formula 1256103)
- vehicle (Placebo Comparator)
  Interventions: Other: vehicle (formula 1256145)
- Reference Octopirox 0.25% (Active Comparator)
  Interventions: Other: reference Octopirox 0.25% (formula 1256149).

INTERVENTIONS:
Other: NaP1%+VitCG3% leave-on lotion (formula 1256103) — leave-on lotion
  Arms: NaP1%+VitCG3% leave-on lotion
Other: vehicle (formula 1256145) — vehicle lotion
  Arms: vehicle
Other: reference Octopirox 0.25% (formula 1256149). — lotion reference Octopirox 0.25%
  Arms: Reference Octopirox 0.25%

SUMMARY:
Edit Brief Summary: To evaluate the NaP lotion effect to decrease dandruff scoring and microbiome rebalance.

Detailed Description: Dandruff is a common scalp disorder affecting almost half of the population of any gender and ethnicity. Skin microflora, in particular Malassezia genus, plays a key etiological role which was demonstrated in many studies.

Malassezia restricta was found as the major fungal species present on the scalps with or without dandruff; while the two main bacterial species found on the scalp surface were Propionibacterium acnes and Staphylococcus epidermidis. Dandruff seems correlated with a higher incidence of Malassezia restricta and Staphylococcus epidermidis and a lower incidence of Cutibacterium acnes.

Also, the link between dandruff and a higher level of scalp surface lipoperoxidation has been recently described. In fact, dandruff scalp surface is also characterized by higher amounts of squalene monohydroperoxide (SQOOH) and malondialdehyde. MDA is a late biomarker derived from sebaceous unsaturated free fatty acids. Some bibliographic elements suggest that these lipid biomarkers could trigger dandruff.

The main objective of that clinical study is to study the effect on dandruff of a leave-on formulation of anti-fungus NaP associated with anti-oxidant VitCG versus vehicle and versus reference leave-on anti-fungus alone Octopirox, all associated with a neutral shampoo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteer;
2. from 18 to 60 years old;
3. Skin Phototype (Fitzpatrick): I to IV;
4. Subject with hair length > 2 cm, and preferentially shorter than shoulder length;
5. Female of childbearing potential, who is not sexually active, or using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study or menopausal woman (with absence of menstruations for less than one year) or post-menopausal woman (with absence of menstruations for more than one year);
6. Subject exhibiting moderate to severe dandruff status of scalp at screening, pre-inclusion and inclusion visit;
7. Subject having at inclusion visit Day 0:

   1. total dandruff score (adherent + non-adherent) > or = 4.5 (ranging from 0 to 10);
   2. adherent dandruff score > or = 2.5 (ranging from 0 to 5);
   3. no limit for non-adherent dandruff score (ranging from 0 to 5);
8. Subject usually using a shampoo 3 times/week and willing to have two to three times/week shampoos during the course of the study;
9. Subject agreeing to use only the supplied products during all the study;
10. Subjects agreeing to have 1 zone of less than 2x2cm2 on the scalp for non-invasive sample taking (swabs);
11. Subject agreeing to have hair shaved on 1 identified zone (1x0.5cm shaved on the high corner of each zone sampling);
12. Subject who demonstrate understanding of the study and willingness to participate as evidenced by voluntary written informed consent and have received a signed and dated copy of the informed consent form.
13. Subject affiliated to a social security or insurance system;
14. Subject willing to comply to the study requirements;
15. Subject who is willing not to take part in another clinical study in another investigating center;
16. Subject who agree to give accurate personal in personal information;
17. Subject who are able to attend all study visits. * The effective contraceptive methods: sexually active female of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide, intravaginal device, intrauterine device (IUD), condom with spermicide.

Exclusion Criteria:

Edit

Eligibility Criteria: Inclusions criterias:

1. Healthy male or female volunteer;
2. from 18 to 60 years old;
3. Skin Phototype (Fitzpatrick): I to IV;
4. Subject with hair length > 2 cm, and preferentially shorter than shoulder length;
5. Female of childbearing potential, who is not sexually active, or using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study or menopausal woman (with absence of menstruations for less than one year) or post-menopausal woman (with absence of menstruations for more than one year);
6. Subject exhibiting moderate to severe dandruff status of scalp at screening, pre-inclusion and inclusion visit;
7. Subject having at inclusion visit Day 0:

   1. total dandruff score (adherent + non-adherent) > or = 4.5 (ranging from 0 to 10);
   2. adherent dandruff score > or = 2.5 (ranging from 0 to 5);
   3. no limit for non-adherent dandruff score (ranging from 0 to 5);
8. Subject usually using a shampoo 3 times/week and willing to have two to three times/week shampoos during the course of the study;
9. Subject agreeing to use only the supplied products during all the study;
10. Subjects agreeing to have 1 zone of less than 2x2cm2 on the scalp for non-invasive sample taking (swabs);
11. Subject agreeing to have hair shaved on 1 identified zone (1x0.5cm shaved on the high corner of each zone sampling);
12. Subject who demonstrate understanding of the study and willingness to participate as evidenced by voluntary written informed consent and have received a signed and dated copy of the informed consent form.
13. Subject affiliated to a social security or insurance system;
14. Subject willing to comply to the study requirements;
15. Subject who is willing not to take part in another clinical study in another investigating center;
16. Subject who agree to give accurate personal in personal information;
17. Subject who are able to attend all study visits. * The effective contraceptive methods: sexually active female of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide, intravaginal device, intrauterine device (IUD), condom with spermicide.

Non-inclusion criterias:

1. Subject with any systemic disorder or skin or scalp disease that would, in the investigator's judgment, significantly affect the interpretation of the study results (e.g. seborrheic dermatitis which shows the syndrome of invasion plaque and/or pityriasis amiantacea, atopic dermatitis, eczema or psoriasis);
2. Female subject who is known to be pregnant or who is intending to become pregnant over the duration of the study;
3. Female subject who is currently breast-feeding or have been breast-feeding in the 6 months prior to the start of the study;
4. Male subject with alopecia grade ≥ V according to Hamilton-Norwood patterns, female subject with alopecia grade I, II or III according to Ludwig patterns (Appendix 3);
5. Subject with frizzy hair influencing the scoring of dandruff;
6. Subject with significant white hair influencing the scoring of dandruff;
7. Subject who has skin marks on the scalp that could interfere with the assessments (e.g. pigmentation, tattoo, scarring etc.);
8. Subject who has used products for the scalp (dyeing, bleaching, permanent waving and straightening …) within the three weeks prior to the study;
9. Subject who has used anti-dandruff treatment (per os or topical) during the last three weeks before the start of the study;
10. Subject who has used cosmetic anti-hair loss treatment (per os or topical) during the last three months before the start of the study, or/and subject who has used medical anti-hair loss treatment (per os or topical, ex: Minoxidil, finasteride, etc…) during the last six months before the start of the study;
11. Subject with personal history of allergy and/or particular reactivity to antidandruff products, and/or to cosmetic products containing tensioactive agents (soaps, shower gel, conditioner …), and/or to latex;
12. Subject who has taken any systemic drug containing corticoids, or anti-fungal, or antibiotics, or any prolonged use of topical drug containing corticoids, or anti-fungal, or antibiotics, or any prolonged use of non-steroidal anti-inflammatory, or anti-histaminic within one month prior to the study;
13. Subject who has taken retinoic acid since less than three months prior to the study;
14. Subject receiving other medication which, in the opinion of the investigator, will affect either the scientific validity of the study or the subject's wellbeing.
15. Subject with a history of medical/surgical events (or surgical events planned) which, in the opinion of the investigator, will affect either the scientific validity of the study or the subject's wellbeing;
16. Immunosuppressed subject;
17. Subject with medical history of skin cancer;
18. Subject who has started, stopped or changed his/her hormonal treatment (including contraceptive pill) in the previous one month prior to the study;
19. Subject practicing regularly water sports and/or having sauna sessions;
20. Subject exposed to the sun or UV rays in an excessive way during the last month prior to the study (according to the investigator);
21. Subject deprived of liberty by adjunction or by official decision;
22. Subject who is participating or who has participated to a clinical study for which the exclusion period is not finished;
23. Subject unable to be contacted by phone;
24. Subject belonging to the staff of the investigating center.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Global score of dandruff status of the scalp: evaluation of adherent and non-adherent dandruff according | Day 0 and Day 28
  scale ranging from 0 (no dandruff) to 5 (maximum score of dandruff adherent and non adherent)

SECONDARY OUTCOMES:
Analysis of Malassezia sp, Cutibacterium sp and Staphylococcus sp | Day 0 and Day 28
  qPCR Malassezia sp, Cutibacterium sp and Staphylococcus sp

CONTACTS AND LOCATIONS:
Locations (1):
- PhD TRIAL, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided